CLINICAL TRIAL: NCT00016783
Title: Intensification of HIV-Specific CD4 and CD8 Activity by Cycling Highly Active Antiretroviral Therapy (HAART) in Pediatric/Adolescent Patients With Less Than 50 HIV RNA Copies/ml
Brief Title: Stopping and Restarting Anti-HIV Drugs in Children and Adolescents With Low Blood Levels of HIV
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: P1015; PACTG P1015; ACTG P1015; 11650 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2001-06-02; First posted 2001-08-31 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Drug Administration Schedule; HIV Protease Inhibitors; CD4 Lymphocyte Count; CD8-Positive T-Lymphocytes; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Antiretroviral Therapy, Highly Active; Treatment Experienced; Treatment Interruption
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Some patients taking anti-HIV drugs as part of highly active antiretroviral therapy (HAART) do not show any HIV in the blood; however, some HIV will remain hidden in the body and, if the drugs are stopped, will return to the blood. The purpose of this study is to determine if short periods of stopping HAART increase the activity of CD8 and CD4 cells (cells of the immune system that fight infection), if repeated stopping of these drugs for longer periods of time and restarting them will increase effectiveness of HAART, and if the increased immune system activity as a result of stopping treatment leads to lower levels of HIV over time.

DETAILED DESCRIPTION:
Some HIV infected patients taking HAART have been able to achieve prolonged suppression of HIV viral load for extended periods of time. However, discontinuing HAART has consistently resulted in HIV's return to plasma. Both CD8 and CD4 cells are markedly reduced in individuals with prolonged HIV suppression; control of and response to cell-associated HIV is dependent on immune-mediated mechanisms involving these cells. It is hypothesized that a brief and low-level increase in HIV levels resulting from HAART interruption might boost HIV-specific CD8 and CD4 T-cell counts. After suppression of viral load with the reintroduction of HAART, the expanded CD8 population might be able to better control viral replication and better respond to cell-associated HIV. Future treatment interruption may lead to longer periods of undetectable viral loads.

Patients are divided into 2 age cohorts, with Cohort 1 consisting of children and adolescents 4 years and older up to 21 years of age, and Cohort 2 consisting of children and adolescents 2 years and older up to 4 years of age. Patients will be assigned to one of 2 groups. Group A patients will participate in drug holiday cycles from HAART and then back to HAART; Group B is a control group that remains on continuous HAART throughout the study. Cycle 1 for Group A patients begins with 18 days of HAART and a 3-day drug holiday. At the end of the drug holiday, viral load is measured and HAART is resumed for 28 days (detectable virus cycle) if viral load is detectable after the drug holiday. If viral load remains below the level of detection, the patient begins the next drug holiday cycle. With each subsequent drug holiday cycle, time off HAART will increase by 2 days. Patients failing 4 repeated detectable virus (28-day treatment) cycles will be taken off study.

Patients will be enrolled in this study for a minimum of 142 weeks. For Group A, HIV viral load and CD4 cell count are measured at the end of each drug holiday and each HAART resumption; HIV-specific CD4 and CD8 responses are measured every 3 cycles; and cell-associated HIV is assessed at entry, at 12-week intervals, and at the end of the study. For Group B, physical exams are conducted and HIV viral load and other blood work are measured every 12 weeks.

ELIGIBILITY:
Note: A Study Monitoring Committee (SMC) recommended on 06/22/05 that this study close, because the primary objectives in this proof-of-concept study could not be achieved. As of 06/28/05, Group A participants will discontinue their drug holiday cycles and will be given the best possible therapy. All participants in this study will have a final study visit to be scheduled as soon as possible, prior to 07/29/05.

Inclusion Criteria:

* HIV infected
* For Cohort 1, CD4 T-cell percent greater than 20
* For Cohort 2, CD4 T-cell percent greater than 25
* Viral load less than 400 copies/ml in the year prior to study entry and less than 50 copies/ml at screening
* Taking anti-HIV drugs (including at least 1 protease inhibitor) and have been on anti-HIV drugs for at least 1 year prior to study entry
* Have been on their current drug regimen for at least 4 months
* Willing to follow study procedures
* Parental or guardian consent if under 18 years old
* Acceptable forms of contraception

Exclusion Criteria:

* Taking abacavir, nevirapine, efavirenz, or delavirdine
* AIDS-related or other infections needing drug treatment at study entry
* Pregnant or breastfeeding
* Have, or have had in the past, diseases (other than HIV infection) or other conditions that, in the doctor's opinion, would interfere with the study
* Taking experimental drugs without the consent of the protocol team

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39
Dates: Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Borkowsky, MD, Study Chair — New York University Medical Center, Pediatric Infectious Diseases
Locations (17):
- United States (16):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Children's Hosp of Denver, Denver, Colorado
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Miami (Pediatric), Miami, Florida
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - St. Lukes/Roosevelt Hosp Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
- San Juan City Hosp, San Juan, Puerto Rico

REFERENCES:
- [Background] Chun TW, Davey RT Jr, Engel D, Lane HC, Fauci AS. Re-emergence of HIV after stopping therapy. Nature. 1999 Oct 28;401(6756):874-5. doi: 10.1038/44755. No abstract available. PMID 10553903
- [Background] Davey RT Jr, Bhat N, Yoder C, Chun TW, Metcalf JA, Dewar R, Natarajan V, Lempicki RA, Adelsberger JW, Miller KD, Kovacs JA, Polis MA, Walker RE, Falloon J, Masur H, Gee D, Baseler M, Dimitrov DS, Fauci AS, Lane HC. HIV-1 and T cell dynamics after interruption of highly active antiretroviral therapy (HAART) in patients with a history of sustained viral suppression. Proc Natl Acad Sci U S A. 1999 Dec 21;96(26):15109-14. doi: 10.1073/pnas.96.26.15109. PMID 10611346
- [Background] Garcia F, Plana M, Vidal C, Cruceta A, O'Brien WA, Pantaleo G, Pumarola T, Gallart T, Miro JM, Gatell JM. Dynamics of viral load rebound and immunological changes after stopping effective antiretroviral therapy. AIDS. 1999 Jul 30;13(11):F79-86. doi: 10.1097/00002030-199907300-00002. PMID 10449278
- [Background] Neumann AU, Tubiana R, Calvez V, Robert C, Li TS, Agut H, Autran B, Katlama C. HIV-1 rebound during interruption of highly active antiretroviral therapy has no deleterious effect on reinitiated treatment. Comet Study Group. AIDS. 1999 Apr 16;13(6):677-83. doi: 10.1097/00002030-199904160-00008. PMID 10397562
- [Background] Ruiz L, Martinez-Picado J, Romeu J, Paredes R, Zayat MK, Marfil S, Negredo E, Sirera G, Tural C, Clotet B. Structured treatment interruption in chronically HIV-1 infected patients after long-term viral suppression. AIDS. 2000 Mar 10;14(4):397-403. doi: 10.1097/00002030-200003100-00013. PMID 10770542